CLINICAL TRIAL: NCT04655820
Title: Maternal and Infant Health and Breast Milk Study in South China
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Huilian Zhu, Professor, Sun Yat-sen University
Other Study IDs: HM-2020
Record Dates: First submitted 2020-11-01; First posted 2020-12-07 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples and breast milk samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study was to investigate the nutrients in breast milk of Chinese mothers and its related factors, as well as exploring the early development of infants.

DETAILED DESCRIPTION:
Breast milk contains a variety of nutrients that are beneficial to the early development of infants, such as lipids, Vitamins and so on. At present, the level of these nutrients in milk and infant formula are lower and which are present in a different form from that in breast milk. Therefore, this study was designed to investigate the level of nutrients in breast milk of Chinese mothers and learn about its related factors, as well as exploring the relationships between these nutrients and the early development of infants.

ELIGIBILITY:
Inclusion Criteria:

* age 20-45 years
* natural delivery, singleton pregnancy
* healthy term infants（at 37-42 weeks of pregnancy）
* don't smoke and drink
* self-evaluation as physical health
* breastfeeding at least until three months of age
* Apgar score > 8
* sign informed consent

Exclusion Criteria:

* suffering from mastitis
* gestational diabetes, hypertension and other metabolic diseases
* AIDS, tuberculosis and other acute or chronic infectious diseases
* severe heart and kidney diseases
* mental system diseases
* cancer and other malignant consumptive disease
* take drugs that affect nutrient metabolism
* infants with congenital and genetic diseases
* with lactation contraindications
* don't agree to sign informed consent

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women and breast-feeding mothers of this study were recruited from Clifford Hospital during the perinatal period or lactation period
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
The level of nutrients in breast milk samples | 14 months
  The nutrients were detected from breast milk samples of mothers by chemical analysis
The level of nutrients in blood samples | 14 months
  The nutrients were detected from blood samples of mothers and infants by chemical analysis

SECONDARY OUTCOMES:
General demographic materials | 14 months
  The general demographic materials of mothers were obtained by questionnaire or medical treatment records
Dietary and lifestyle information | 14 months
  Dietary and lifestyle information of mothers were obtained by Food Frequency Questionnaire and 24-hour meal review questionnaire
Health follow-up | 14 months
  Dietary and health outcome of infants were obtained by questionnaire or medical treatment records

CONTACTS AND LOCATIONS:
Locations (1):
- SunYat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No